CLINICAL TRIAL: NCT03684811
Title: A Phase 1b/2 Study of FT-2102 in Patients With Advanced Solid Tumors and Gliomas With an IDH1 Mutation
Brief Title: A Study of FT-2102 in Patients With Advanced Solid Tumors and Gliomas With an IDH1 Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2102-ONC-102
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cohort 1a and 1b: Glioma (Advanced Gliomas and Glioblastoma Multiforme); Cohort 2a and 2b: Hepatobiliary Tumors (Hepatocellular Carcinoma, Bile Duct Carcinoma, Intrahepatic Cholangiocarcinoma, Other Hepatobiliary Carcinomas); Cohort 3a and 3b: Chondrosarcoma; Cohort 4a and 4b: Intrahepatic Cholangiocarcinoma; Cohort 5a: Other Non-Central Nervous System Solid Tumors With IDH1 Mutations
Keywords: Olutasidenib
MeSH Terms: conditions — Glioblastoma; Carcinoma, Hepatocellular; Bile Duct Neoplasms; Cholangiocarcinoma | interventions — olutasidenib; Azacitidine; Nivolumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1b Dose Confirmation Single Agent (Cohorts 1a-5a) (Experimental)
  Interventions: Drug: FT-2102
- Phase 2 Cohorts FT-2102 Single Agent (Cohorts 1a-5a) (Experimental)
  Interventions: Drug: FT-2102
- Phase 1b and 2 Cohorts Combination (Cohorts 1b and 3b) (Experimental)
  Interventions: Drug: FT-2102; Drug: Azacitidine
- Phase 1b and 2 Cohort Combination (Cohort 2b) (Experimental)
  Interventions: Drug: FT-2102; Biological: Nivolumab
- Phase 1b and 2 Cohort Combination (Cohort 4b) (Experimental)
  Interventions: Drug: FT-2102; Drug: Gemcitabine and Cisplatin

INTERVENTIONS:
Drug: FT-2102 — FT-2102 will be supplied as a 150 mg capsule and will be administered per the protocol defined frequency and dose level.
Drug: Azacitidine — Azacitidine will be administered per the site's standard of care.
  Other Names: Vidaza
  Arms: Phase 1b and 2 Cohorts Combination (Cohorts 1b and 3b)
Biological: Nivolumab — Nivolumab will be administered per the site's standard of care.
  Other Names: Opdivo
  Arms: Phase 1b and 2 Cohort Combination (Cohort 2b)
Drug: Gemcitabine and Cisplatin — Gemcitabine and cisplatin will be administered per the site's standard of care.
  Other Names: Gemzar and Platinol
  Arms: Phase 1b and 2 Cohort Combination (Cohort 4b)

SUMMARY:
This Phase 1/2 study will evaluate the safety, efficacy, PK, and PD of FT-2102 as a single agent and in combination with other anti-cancer drugs in patients with advanced solid tumors and gliomas.

The study is divided into two parts: single agent FT-2102 followed by combination therapy.

Part 1: A single agent, open-label study in up to five cohorts (glioma, hepatobiliary tumors, chondrosarcoma, intrahepatic cholangiocarcinoma, and other IDH1 mutant solid tumors) that will include a Phase 1 dose confirmation followed by a Phase 2 investigation of clinical activity in up to 4 cohorts. During the dose confirmation, additional doses or altered dose schedules may be explored.

Part 2: An open-label study of FT-2102 in combination with other anti-cancer agents. Patients will be enrolled across 4 different disease cohorts, examining the effect of FT-2102 + azacitidine (glioma and chondrosarcoma), FT-2102 + nivolumab (hepatobiliary tumors), and FT-2102 + gemcitabine/cisplatin (intrahepatic cholangiocarcinoma). There will be a safety lead-in followed by a Phase 2 evaluation in up to four cohorts of patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have documented IDH1-R132 gene-mutated disease as evaluated by site
* Glioma: Advanced glioma that has recurred or progressed following standard therapy, or that has not responded to standard therapy.
* Hepatobiliary cancer that is relapsed/refractory or intolerant to approved standard-of-care therapy (including: hepatocellular carcinoma, bile duct carcinoma, intrahepatic cholangiocarcinoma or other hepatobiliary carcinomas)
* Chondrosarcoma that is relapsed or refractory and either locally advanced or metastatic and not amenable to complete surgical excision
* Intrahepatic cholangiocarcinoma that is advanced nonresectable or metastatic cholangiocarcinoma not eligible for curative resection or transplantation. Phase 1b/Safety Lead-in of Phase 2: relapsed or refractory disease. Combination Phase 2 (beyond Safety Lead-in): have received no more than 1 cycle of gemcitabine/cisplatin therapy
* Other solid tumors that have relapsed or refractory to standard-of-care therapy with no other available therapeutic options
* Good performance status
* Good kidney and liver function

Key Exclusion Criteria:

* Prior solid organ or hematopoietic cell transplant
* Prior treatment with IDH1 inhibitor (single agent cohorts only)
* Congestive heart failure (New York Heart Association Class III or IV) or unstable angina pectoris. Previous history of myocardial infarction within 1 year prior to study entry, uncontrolled hypertension or uncontrolled arrhythmias
* Unstable or severe, uncontrolled medical condition (e.g., unstable cardiac function, unstable pulmonary condition, including pneumonitis and/or interstitial lung disease, and uncontrolled diabetes)
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* PD-1 only: active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barrett, Study Director — Forma Therapeutics
Locations (26):
- United States (14):
  - Banner MD Anderson, Gilbert, Arizona
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa, Holden Comprehensive Cancer Institute, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Baylor Scott and White Medical Center, Temple, Texas
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - Medical College of Wisconsin, Froedtert Hospital, Milwaukee, Wisconsin
- Australia (2):
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne
- France (4):
  - Centre de Lutte Contre Cancer (CLCC) - Institute Bergonie, Bordeaux
  - Centre de Lutte Cancre (CLCC) - Lyon, Lyon
  - Hospital de la Timone, Marseille
  - Institut Gustave Roussy Cancer Campus, Villejuif
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Vall D'Hebron University Hospital, Barcelona, Spain
- United Kingdom (2):
  - Cancer Research Beatson Institute, Glasgow
  - The Royal Marsden Hospital, London

REFERENCES:
- [Derived] Jones RL, Groisberg R, Blay JY, Colman H, De La Fuente M, Roxburgh P, Chao MM, Tian H, Duffaud F, Bahleda R, Van Tine BA. Olutasidenib in recurrent/relapsed locally advanced or metastatic IDH1-mutated chondrosarcoma: phase 1b/2 trial. Nat Commun. 2026 Jan 29. doi: 10.1038/s41467-026-68716-6. Online ahead of print. PMID 41611702

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1A: Glioma
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
- Cohort 1B: Glioma
  Olutasidenib (150 QD or 150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
  Azacitidine (75 mg/m2/day × 7 days every 28 days) was administered intravenously (or subcutaneously) daily for 7 days in combination with olutasidenib.
- Cohort 2A: Hepatobiliary Tumors (Hepatocellular Carcinoma, Bile Duct Carcinoma, Intrahepatic Cholangiocarcinoma, Other Hepatobiliary Carcinomas)
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
- Cohort 2B: Hepatobiliary Tumors (Hepatocellular Carcinoma, Bile Duct Carcinoma, Intrahepatic Cholangiocarcinoma, Other Hepatobiliary Carcinomas)
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
  Nivolumab (240 mg intravenously every 2 weeks) was to be administered in combination with olutasidenib.
  No patients were enrolled into Cohort 2b.
- Cohort 3A: Chondrosarcoma
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
- Cohort 3B: Chondrosarcoma
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
  Azacitidine (75 mg/m2/day × 7 days every 28 days) was to be administered intravenously (or subcutaneously) daily for 7 days in combination with olutasidenib.
  No patients were enrolled in Cohort 3b.
- Cohort 4A: Intrahepatic Cholangiocarcinoma
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
- Cohort 4B: Intrahepatic Cholangiocarcinoma
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
  GemCis (cisplatin [25 mg/m2] followed by gemcitabine [1000 mg/m2], each administered on Days 1 and 8, every 3 weeks, for 8 cycles of up to 24 weeks) was to be administered in combination with olutasidenib.
  No patients were enrolled in Cohort 4b.
- Cohort 5A: Other Non-Central Nervous System Solid Tumors With IDH1 Mutations
  Olutasidenib (150 mg BID) was administered orally in continuous 28 day cycles until criteria for treatment discontinuation were met.
Period: Overall Study
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 2B | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Cohort 5A
Started | 26 | 6 | 8 | 0 | 23 | 0 | 24 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 26 | 6 | 8 | 0 | 23 | 0 | 24 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set - Patients who have received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A | Total
Number analyzed (Participants) | 26 | 6 | 8 | 23 | 24 | 6 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (9.13) | 42.0 (7.21) | 59.9 (10.47) | 55.1 (10.68) | 57.1 (12.56) | 61.3 (18.3) | 52.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 6 | 6 | 17 | 4 | 44
  Male | 17 | 4 | 2 | 17 | 7 | 2 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 2 | 2 | 0 | 7
  Not Hispanic or Latino | 22 | 5 | 5 | 15 | 16 | 4 | 67
  Unknown or Not Reported | 2 | 0 | 3 | 6 | 6 | 2 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 25 | 6 | 3 | 17 | 17 | 3 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 6 | 5 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: DLTs are AEs unrelated to the underlying disease and considered related to FT-2102. For non-hematologic AEs: Grade 3 or higher per CTCAE v 4.03 criteria except Grade 3 nausea, vomiting, diarrhea, or rash: lasting <72 hours (with optimal medical management) or clinically relevant Grade 3 or higher non-hematologic laboratory finding. For hematologic AEs: Grade 3 or higher thrombocytopenia or febrile neutropenia or Grade 4 or higher neutropenia lasting for >7 days.
Time Frame: Day 1-28
Population: All patients in the Safety Lead-in Period who either experienced a DLT during Cycle 1 or completed at least 75% of the prescribed Cycle 1 dose. The Safety-Lead-in Period will employ a traditional 3+3 design, whereby 3 patients with any of the solid tumors (Cohorts 2a-5) and 3 patients with gliomas (Cohort 1a) are treated with FT-2102 150 mg BID and monitored for DLTs during the first cycle of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B | Cohort 3A | Cohort 5A
Number analyzed (Participants) | 3 | 5 | 3 | 1
Participants | 0 | 2 | 0 | 1

2. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) as per RANO (2010) criteria for patients with high grade glioma (Cohorts 1a and 1b). For patients with low grade glioma, ORR is defined as CR+PR+minor response (MR) as per LGG RANO criteria (2011). For Cohorts 2-5, ORR is defined as CR+PR as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Time Frame: While on treatment
Population: The Response-Evaluable Analysis Set is defined as all patients with measurable disease at baseline are included in the Safety Analysis Set and had at least 1 post-baseline response assessment or discontinued the treatment phase due to disease progression (including death caused by disease progression) within 8 weeks (+2-week window) of the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 25 | 5 | 8 | 21 | 19 | 6
Participants | 2 | 0 | 1 | 0 | 0 | 0

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Area under the plasma concentration versus time curve (AUC) summarized for Cycle 1 and Cycle 2
Time Frame: Cycles 1: Day 1 (0, 1, 2, 4, 8 hours post dose), Days 2, 8, 15, 22 pre dose. Cycles 2 Day 1 (0, 1, 2, 4, 8 hours post dose).
Population: The PK analysis set is defined as patients from Stage 1 who have received at least one dose of FT-2102 and for whom it is possible to calculate at least one primary PK parameter (e.g. Cmax, AUC).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 9 | 6 | 8 | 9 | 12 | 5
h*ng/mL
  Cycle 1: number analyzed (Participants) | 9 | 6 | 8 | 9 | 11 | 4
  Cycle 1 | 6840 (3062.9) | 6190 (2113.0) | 13140 (6018.9) | 12000 (2907.1) | 10780 (6379.1) | 11030 (6781.6)
  Cycle 2: number analyzed (Participants) | 8 | 3 | 6 | 8 | 8 | 4
  Cycle 2 | 20390 (5975.5) | 21210 (5775.0) | 27580 (4531.3) | 28170 (9052.5) | 24400 (8663.1) | 39540 (12573)

4. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Peak Plasma Concentration (Cmax) was summarized for Cycle 1 and Cycle 2.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 9 | 6 | 8 | 9 | 12 | 5
ng / mL
  Cycle 1: number analyzed (Participants) | 9 | 6 | 8 | 9 | 11 | 5
  Cycle 1 | 388.1 (154.92) | 369.5 (127.84) | 879.4 (432.37) | 863.4 (313.71) | 744.1 (526.73) | 815.4 (432.32)
  Cycle 2: number analyzed (Participants) | 8 | 3 | 6 | 8 | 8 | 4
  Cycle 2 | 2965 (917.89) | 2870 (540.28) | 4045 (527.02) | 4104 (1326.0) | 3650 (985.06) | 5663 (1897.8)

5. Secondary Outcome: Time of Peak Plasma Concentration (Tmax)
Description: Time of peak plasma concentration (Tmax) was summarized for Cycle 1 and Cycle 2.
Time Frame: as for outcome 3
Population: The PK analysis set is defined as patients who have received at least one dose of FT-2102 and for whom it is possible to calculate at least one primary PK parameter (e.g. Cmax, AUC).
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 9 | 6 | 8 | 9 | 12 | 5
hours
  Cycle 1: number analyzed (Participants) | 9 | 6 | 8 | 9 | 11 | 5
  Cycle 1 | 4.18 [1.95 to 20.25] | 3.95 [1.92 to 27.23] | 15.27 [2.03 to 24.33] | 16.37 [1.02 to 23.92] | 7.50 [1.00 to 24.00] | 4.17 [1.00 to 23.05]
  Cycle 2: number analyzed (Participants) | 8 | 3 | 6 | 8 | 8 | 4
  Cycle 2 | 1.97 [0.00 to 7.57] | 4.00 [3.97 to 4.05] | 1.05 [1.00 to 7.85] | 1.98 [0.95 to 4.00] | 1.04 [0.00 to 4.22] | 1.52 [0.00 to 7.58]

6. Secondary Outcome: Time for Half of the Drug to be Absent in Blood Stream Following Dose (T 1/2)
Description: Time for half of the drug to be absent in blood stream following dose (T 1/2)
Time Frame: as for outcome 3
Population: The PK analysis set is defined as patients who have received at least one dose of FT-2102 and for whom it is possible to calculate at least one primary PK parameter (e.g. Cmax, AUC). Results were not estimable for this outcome measure because of the limited sampling interval post Day 1.
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 9 | 6 | 8 | 8 | 11 | 4
ng / mL | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1.

7. Secondary Outcome: Apparent Clearance (CL/F)
Description: Rate at which drug is removed from the blood stream (CL/F).
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: units
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 9 | 6 | 8 | 8 | 11 | 4
units | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA (NA) — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1.

8. Secondary Outcome: Rate of Drug Distribution Within the Blood Stream (Vd/F)
Description: Rate of drug distribution within the blood stream (Vd/F)
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number; unit: units
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 9 | 6 | 8 | 8 | 11 | 4
units | NA — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1. | NA — Results were not estimable for this outcome measure because of the limited sampling interval post Day 1.

9. Secondary Outcome: Olutasidenib Concentration Within Cerebro-spinal Fluid (CSF)
Description: Olutasidenib concentration within CSF (Glioma Cohorts 1-A and 1-B only). Due to sparse data, analysis was not conducted by timepoint.
Time Frame: CSF sample for drug concentration was collected at Day 1 of Cycles 1 and 3 (each cycle is 28 days) and through study completion, up to 24 weeks, on average.
Population: Glioma patients who had a CSF sample obtained while on study treatment were analyzed. CSF samples were not collected for cohorts 2-5, per protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 2 | 0
ng/mL | 27.15 (6.57) |

10. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival from time of entry on study. Progression-free survival (PFS) is defined as the time from the first dose to disease progression as determined by applicable disease criteria or death due to any cause, whichever was sooner. Disease progression as measured by the appropriate response criteria, unless deemed by the Investigator to be receiving clinical benefit
Time Frame: From time of entry on study through progression, up to 24 weeks, on average
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 25 | 5 | 8 | 21 | 19 | 6
weeks | 8.21 [7.14 to 37.50] | 8.29 [8.14 to 9.43] | NA [7.00 to NA] — Median not reached | 8.57 [7.43 to 22.14] | 8.29 [7.00 to 17.71] | 8.07 [7.57 to 31.00]

11. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time (in weeks) from start of treatment until disease specified progression.
Time Frame: From first dose of study drug through time of disease progression
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 25 | 5 | 8 | 21 | 19 | 6
weeks | 8.21 [7.14 to 37.50] | 8.29 [8.14 to 9.43] | NA [7.0 to NA] — Median not reached | 15.00 [7.43 to 24.00] | 13.86 [7.29 to 24.14] | 8.14 [8.00 to 31.00]

12. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR), defined as the time from the first response to documented disease progression as determined by applicable disease criteria. First response is defined as first observation of overall response of CR+PR+MR (glioma) or CR+PR (Cohort 2-5). Disease progression as measured by the appropriate response criteria, unless deemed by the Investigator to be receiving clinical benefit
Time Frame: From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 44 weeks
Population: Response-Evaluable Analysis Set defined as all patients with measurable disease at baseline are included in the Safety Analysis Set and had at least 1 post-baseline response assessment or discontinued the treatment phase due to disease progression (including death caused by disease progression) within 8 weeks (+2-week window) of the first dose of study treatment. Duration of response was calculated on the subset of patients in the Response Evaluable Set who experienced an Overall Response.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 0
weeks | 43.71 [43.71 to 43.71] |  | NA [NA to NA] — Median Not Reached |  |  |

13. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS), defined as the time in weeks from the first dose to death due to any cause or date last known alive at end of follow-up
Time Frame: From date of first dose until the date of death from any cause, assessed up to 101 weeks
Population: Safety Analysis Set - Patients who have received at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 26 | 6 | 8 | 23 | 24 | 6
weeks | 75.00 [45.86 to NA] — Upper Quartile not estimable due to number of censored patients | NA [NA to NA] — Median Not Reached due to number of censored patients | NA [32.00 to NA] — Median Not Reached due to number of censored patients | NA [23.14 to NA] — Median Not Reached due to number of censored patients | 36.43 [10.29 to NA] — Upper Quartile not estimable due to number of censored patients | NA [33.71 to NA] — Median Not Reached due to number of censored patients

14. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) in weeks. TTR is defined as the time from first dose to first response. First response is defined as first observation of overall response of CR+PR+MR (glioma) or CR+PR (Cohort 2-5).
Time Frame: Response may be observed from time of first dose through time of treatment discontinuation, up to 2 years.
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 0
weeks | 38.07 [8.29 to 67.86] |  | 31.43 [31.43 to 31.43] |  |  |

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose (Up to approximately 2 years)
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 3A | Cohort 4A | Cohort 5A
All-Cause Mortality (participants affected / at risk) | 2/26 | 0/6 | 0/8 | 2/23 | 4/24 | 1/6
Serious Adverse Events (participants affected / at risk) | 11/26 | 3/6 | 5/8 | 12/23 | 9/24 | 1/6
Other Adverse Events (participants affected / at risk) | 26/26 | 6/6 | 8/8 | 21/23 | 23/24 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A (N=26) | Cohort 1B (N=6) | Cohort 2A (N=8) | Cohort 3A (N=23) | Cohort 4A (N=24) | Cohort 5A (N=6)
Disease Progression (General disorders) | 6 | 1 | 1 | 5 | 6 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A (N=26) | Cohort 1B (N=6) | Cohort 2A (N=8) | Cohort 3A (N=23) | Cohort 4A (N=24) | Cohort 5A (N=6)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 4 | 6 | 15 | 9 | 4
Constipation (Gastrointestinal disorders) | 7 | 2 | 4 | 7 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 1 | 1 | 2 | 5 | 3
Vomiting (Gastrointestinal disorders) | 5 | 1 | 2 | 3 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 13 | 2 | 3 | 7 | 8 | 1
Disease progression (General disorders) | 6 | 1 | 1 | 5 | 6 | 1
Asthenia (General disorders) | 0 | 1 | 2 | 4 | 5 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Candida infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 5 | 3 | 7 | 9 | 4
Aspartate aminotransferase increased (Investigations) | 5 | 4 | 2 | 7 | 11 | 4
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 4 | 6 | 8 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 1 | 6 | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 2 | 2 | 4 | 3 | 0
Red blood cell count decreased (Investigations) | 1 | 1 | 2 | 2 | 4 | 2
Platelet count decreased (Investigations) | 4 | 2 | 0 | 1 | 4 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 3 | 2 | 2
Weight decreased (Investigations) | 2 | 0 | 0 | 4 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 3 | 1 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 2 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 4 | 10 | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 4 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 5 | 1 | 2 | 5 | 1 | 0
Headache (Nervous system disorders) | 8 | 1 | 2 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 2 | 3 | 0 | 0
Seizure (Nervous system disorders) | 5 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 1 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 0 | 0 | 4 | 2 | 1
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 5 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 5 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 0 | 2 | 3 | 1 | 0
Hot flush (Vascular disorders) | 2 | 1 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principle investigators are required to ensure Forma has at least 60 days time for review and to provide input or request modifications where pertinent.

DOCUMENTS (2):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03684811/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03684811/SAP_001.pdf